CLINICAL TRIAL: NCT06225726
Title: Elastographic Analysis of Urothelial Bladder Tumours. Correlation of Elastography With Urodynamic Study and Tumour Grade
Brief Title: Elastographic Analysis of Urothelial Bladder Tumours
Acronym: SONURO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR230158 - SONURO
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Elastographic Measurement; Intravesical Pressure Measurement
Keywords: urothelial bladder tumours; tumour grade; ShearWave Elasticity; Urodynamic study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental : Urothelial bladder tumour: Patient with an indication of transurethral resection of the bladder. Following the Urology consultation, the patient will be called for a trans-urethral bladder resection within 1 month. The patient will be admitted to the Urology Department of the Tours University Hospital the previous day.
  Interventions: Procedure: urethral bladder resection

INTERVENTIONS:
Procedure: urethral bladder resection — urethral bladder resection. Per-operative bladder ultrasound elastography and simultaneous cystometry

SUMMARY:
The preoperative evaluation of bladder tumors includes either computed tomography, magnetic resonance imaging in B-mode, or a cystoscopy in the absence of a radiological diagnosis. The diagnosis is confirmed after a transurethral resection of the bladder (TURB) and a histopathological analysis.

Ultrasound is a non-invasive imaging technique that uses high-frequency sound waves to produce images of internal structures. Conventional ultrasound in B-mode can only provide details about the tumor's number, size, and location.

Elastography uses ultrasound imaging techniques to examine the stiffness of a tissue. Using the Aixplorer system many recently published papers suggested that ShearWave Elasticity (SWE) imaging, enables the differentiation of low- from high-grade breast tumors by assessing the elasticity of the tissue.

Investigators intend to evaluate the stiffness of bladder tumors with ultrasound elastography in comparison with cystometry parameters and tumoral grade.

DETAILED DESCRIPTION:
According to European and French guidelines, Transurethral resection of the bladder can be followed by an administration of early postoperative intravesical chemotherapy. This treatment is indicated in the absence of presumed high grade tumor (preoperative high grade cytology) and in the absence of post-operative haematuria and bladder perforation. Unfortunately, urine cytology has a sensitivity for the detection of high-grade tumour of only 50%. Therefore, it is essential to predict more precisely the bladder tumor grade.

Ultrasound is a non-invasive imaging technique that uses high-frequency sound waves to produce images of internal structures. Conventional ultrasound in B-mode can only provide details about the tumor's number, size, and location.

Elastography uses ultrasound imaging techniques to examine the stiffness of a tissue. Using the Aixplorer system many recently published papers suggested that ShearWave Elasticity (SWE) imaging, enables the differentiation of low- from high-grade breast tumors by assessing the elasticity of the tissue. Many studies have shown a significant correlation between ultrasound elastography of the bladder wall with measurements of the detrusor pressure. Only one study, conducted by Huang et al., have assessed its application in the evaluation of bladder cancer with an intraluminal transducer. A significant difference between elasticity of low grade and high grade bladder tumors was found. However, no data on the impact of the intravesical volume over the tumoral elasticity is available.

The objective of this project is to evaluate the correlation between the ultrasound Elastography of urothelial bladder tumors with their tumoral grade before transurethral resection of the bladder.

Knowing that ultrasound Elastography is impacted by the pressure applied to a tissue, investigators intend to measure the tumoral elasticity - with an abdominal ultrasound transducer - during bladder filling with a monitoring of the intravesical pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Bladder tumour visualised on abdominal ultrasound or estimated to be more than 2 cm in diameter by fibroscopy or CT scan
* Primary resection

Exclusion Criteria:

* BMI > 30 kg/m2,
* Bladder catheterisation,
* Previous bladder or prostate surgery,
* Previous intravesical instillation (BCG / Ametycine)
* Previous pelvic radiotherapy,
* Person having objected to data processing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a bladder tumour which needs a primary trans-urethral resection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Ultrasound elastography measurements | 10 minutes, during surgery
  Measure of tumoral ultrasound elasticity (in kPa) with an abdominal ultrasound transducer.

SECONDARY OUTCOMES:
Comparison between ultrasound results and histology | through study completion, an average of 10 months
  Histology criteria : tumoral grade according to WHO classification (1973 and 2022)
Comparison between ultrasound results and cystometry | through study completion, an average of 10 months
  Cystometry data using an urodynamic system during the cystoscopy and simultaneous ultrasound measurements at successive filling volumes : intravesical pressure (cmH2O).

CONTACTS AND LOCATIONS:
Overall Officials: Franck BRUYERE, Principal Investigator — University Hospital
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided